CLINICAL TRIAL: NCT06896123
Title: Studio Sulla Fattibilità e Sul Potenziale Riabilitativo Dell'Esperienza Artistica di Dance Well Nei Pazienti Affetti da Malattia di Parkinson
Brief Title: Dance Well Therapy: a Study for Evaluating Efficacy, Safety, and Feasibility
Acronym: DWpsVMF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Casa di Cura Villa Margherita Fresco (Other)
Responsible Party: Principal Investigator, Giampietro Rupolo, President of KOS Medical Group, Casa di Cura Villa Margherita Fresco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DWpsVMF
Record Dates: First submitted 2025-03-10; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: PD; Dance Well; Rehabilitation Therapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DanceWell Group (Experimental): 12 PD patients underwent 4-week Dance Well Program
  Interventions: Behavioral: Dance Well: an artistic, multisensory dance intervention based on art and music
- Conventional Therapy Group (Active Comparator): 12 PD patients underwent 4-week Conventional Therapy Program
  Interventions: Behavioral: Conventional motor therapy group

INTERVENTIONS:
Behavioral: Dance Well: an artistic, multisensory dance intervention based on art and music — DW is specifically designed for people with early to mild severe PD and aims to de-liver multiple stimuli, including rhythmical auditory cues, proprioceptive and sensorimo-tor stimulation, balance training, and aerobic exercise, using carefully selected music to cue movement and promote relaxation. The components of DW are relatively simple and easy to be learned and performed for people with compromised mobility. The intervention is also enjoyable and engaging, as reported for other genres of dance
  Arms: DanceWell Group
Behavioral: Conventional motor therapy group — Conventional Motor Therapy consisted on 60-minute conventional physiotherapy, twice a week, for four weeks
  Arms: Conventional Therapy Group

SUMMARY:
A new and in-teresting complementary approach for rehabilitation of parkinsonian patients is represented by "Dance Well", which is an artistic, multisensory dance intervention based on art and music. This study aims to evaluate the efficacy, feasibility, and safety of a 4-week Dance Well (DW) program in PD patients in early-medium disease stages.

DETAILED DESCRIPTION:
Background/Objectives: Parkinson's disease (PD) is a complex neurodegenerative disorder re-sponsible for both motor and non-motor disturbances impairing the motor behaviour. This com-plexity needs for integrated, multidisciplinary and comprehensive models of care. A new and in-teresting complementary approach is represented by "Dance Well," i.e., an artistic, multisensory dance intervention based on art and music. This pilot study aims to evaluate the efficacy, feasibility, and safety of a 4-week Dance Well (DW) program in PD patients in early-medium disease stages. Methods: Twenty-four PD patients (H&Y ≤ 3; MoCA score ≥ 13.8) were enrolled and randomly allocated into two groups, both with a twice per week frequency and lasting 4 weeks: one group underwent the DW program, while the other underwent conventional physiotherapy (CPT). De-mographic, biometric, and clinical data were collected. To study the treatment effect, motor (Unified PD Rating Scale-III, Timed-up and Go Test, Berg Balance Scale, 6-Minute Walk Test, and Falls Efficacy Scale), cognitive (Corsi Supra Span Test, Trial Making Test A and B-A), and affective (Beck Depression Inventory, State-Trait Anxiety Inventory, Apathy Evaluation Scale) outcome measures were as-sessed, before and after rehabilitation program. To study the treatment compliance and safety, number of dropouts and any adverse events (such as injuries and falls) were recorded.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PD according to the UK Parkinson's Disease Society Brain Bank clinical diagnostic criteria; rate score 0-3 on the modified Hoehn & Yahr (H&Y) scale.

Exclusion Criteria:

* other neurological or psychiatric diseases other than PD;
* serious visual and/or auditory deficits;
* orthopedic-muscular and or co-morbid medical conditions precluding partici-pation in dance;
* cognitive decline (MoCA score < 13,8)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
UPDRS III | Form the enrollment to the end of treatment at 4 weeks
  UPDRS III (Unified Parkinson's Disease Rating Scale, Part III) is a clinical tool used to assess motor function in Parkinson's disease patients. It evaluates symptoms such as tremors, rigidity, bradykinesia, postural stability, gait, and rapid alternating movements. Each item is scored from 0 (no impairment) to 4 (severe impairment), with the total score indicating the overall severity of motor symptoms.

SECONDARY OUTCOMES:
Berg Balance Scale (BBS) | Form the enrollment to the end of treatment at 4 weeks
  The Berg Balance Scale (BBS) is a widely used tool designed to assess static balance and fall risk in adults. Here are the key points. The scale must be administered by a trained physical therapist, and it consists of 14 tasks, each scored on a 5-point scale (0-4), with 0 indicating the lowest level of function and 4 the highest. Tasks includes activities like sitting to standing, standing unsupported, reaching forward, and turning 360 degrees. It typically takes 15-20 minutes to administer.
6-Minute Walk Test (6MWT) | Form the enrollment to the end of treatment at 4 weeks
  The 6-Minute Walk Test (6MWT) is a simple and effective tool used to assess aerobic capacity and endurance, measuring the distance as far as possible an individual can walk in six minutes on a flat, straight surface. The outcome is the total distance walked in meters within the six-minute period. Participants are encouraged to walk back and forth along a marked walkway, with standardized encouragement provided at specific intervals. This test is widely used in clinical and research settings to evaluate walk and to monitor changes over time.
Timed Up and Go (TUG) Test | Form the enrollment to the end of treatment at 4 weeks
  The Timed Up and Go (TUG) Test is a simple and quick assessment used to evaluate mobility, balance, walking ability, and fall risk. It involves the participant sitting in a chair, standing up upon command, walking 3 meters (10 feet), turning around, walking back to the chair, and sitting down. The score consists in time taken to complete the task it is col-lected in seconds. A longer time indicates greater risk of falling.
Corsi Supra-Span Block Tapping Test | Form the enrollment to the end of treatment at 4 weeks
  The Corsi Supra-Span Block Tapping Test aims to assess visuo-spatial working memory and learning processes for a number of information overcoming the short-term memory span. Placed in front of a board, where nine identical blocks have arranged, par-ticipants are required to reproduce a sequence of 9 blocks tapped by the examiner. Partici-pants can learn and recall the sequences through repeated trials, for a maximum of 18 rep-etitions. The global score is the sum of the score obtained for each stem of correct sequence.
Trail Making Test (TMT) A and B-A | Form the enrollment to the end of treatment at 4 weeks
  Trail Making Test (TMT) A is a paper-and-pencil test, aimed to assess visual atten-tion, while TMT B-A score aims to assess task switching. Part A involves connecting 25 numbered circles in ascending order as quickly as possible. The time taken to complete each part is recorded in seconds, representing the score. B-A score represents the subtrac-tion among TMT B and TMT A scores (where, the part B, aimed to evaluate divided atten-tion consists in connecting 25 circles, alternating between numbers and letters - e.g., 1-A-2-B - as quickly as possible). Higher times indicate greater impairment.
Beck Depression Inventory (BDI) | Form the enrollment to the end of treatment at 4 weeks
  Beck Depression Inventory (BDI) is a self-administered questionnaire, aimed to measure the depression symptoms. It consists of 21 Items, each of them item corresponds to a symptom of depression. Each item is rated on a 4-point scale (0-3). The total score ranges from 0 to 63, with higher scores indicating more severe depression.
State-Trait Anxiety Inventory (STAI-I) part I | Form the enrollment to the end of treatment at 4 weeks
  State-Trait Anxiety Inventory (STAI-I) part I is a self-administered questionnaire, aimed to measure state anxiety. It consists of 20 items assessing how one feels at the evalu-ation moment. Each item is rated on a 4-point scale, with higher scores indicating greater anxiety.
Apathy Evaluation Scale (AES) | Form the enrollment to the end of treatment at 4 weeks
  Apathy Evaluation Scale (AES), is a self-administered questionnaire, aimed to meas-ure the level of apathy in individuals. It consists of 18 Items (each of them rated on a 4-point scale), assessing behavioral, cognitive, and emotional aspects of goal-directed be-havior. The total score ranges from 18 to 72, with higher scores indicating greater apathy.

CONTACTS AND LOCATIONS:
Locations (1):
- Fresco Parkinson Center - Villa Margherita (KOS group), Arcugnago, VI, Italy

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data (IPD) due to concerns related to patient privacy and data security. Ensuring the confidentiality and protection of our participants' personal information is a top priority. Additionally, the resources required to anonymize and manage data sharing securely are not available for this study